CLINICAL TRIAL: NCT01893255
Title: A Multi-national, Multi-center Non-interventional Study in Rheumatoid Arthritis (RA) Patients Who Are Treated With Tocilizumab
Brief Title: A Non-Interventional Study in Patients With Rheumatoid Arthritis Who Are Treated With RoActemra/Actemra (Tocilizumab)
Status: Withdrawn | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28443
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the use and efficacy of RoActemra/Actemra (tocilizumab) in monotherapy in routine clinical practice in patients with rheumatoid arthritis. Eligible patients initiated on RoActemra/Actemra treatment according to the approved label will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) ACR criteria
* Patients in whom the treating physician has made the decision to commence RoActemra/Actemra treatment in accordance with the local label; this can include patients who have received RoActemra/Actemra treatment within 8 weeks prior to the enrolment visit
* Patients who for any reason do not take methotrexate and the treating physician has made a decision to prescribe RoActemra/Actemra as monotherapy
* Patients who were previously on a TNF inhibitor as monotherapy, and the treating physician has made a decision to prescribe RoActemra/Actemra as monotherapy
* Concomitant treatment with corticosteroids (orally and intra-articularly) and/or NSAIDs is allowed

Exclusion Criteria:

* Patients who have received RoActemra/Actemra more than 8 weeks prior to the enrolment visit
* Patients who have previously received RoActemra/Actemra in a clinical trial or for compassionate use
* Patients receiving concomitant DMARD treatment for rheumatoid arthritis (e.g. hydroxychloroquine, sulfasalazine, methotrexate, leflunomide, gold compounds, cyclosporine)
* Patients who have received treatment with an investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* Patients with a history of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis initiated on treatment with RoActemra/Actemra in monotherapy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients on RoActemra/Actemra at 6 months after treatment initiation | Month 6

SECONDARY OUTCOMES:
Clinical/demographic patient characteristics at initiation of RoActemra/Actemra treatment | approximately 6 months
Rates of dose modifications/interruptions | approximately 6 months
Efficacy: Response according to total joint count evaluation by DAS28/EULAR/SDAI/CDAI/ACR | approximately 6 months
Physician's Global Assessment of Disease Activity | approximately 6 months
Safety: Incidence of adverse events | approximately 6 months
Patient reported outcomes (Patient Global Assessment of disease activity, HAQ-DI, VAS-Fatigue, severity of pain and morning stiffness) | approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche